CLINICAL TRIAL: NCT03968887
Title: Correlation Between Plasma Oxidized Low Density Lipoprotein Levels And Postoperative Delirium
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-092
Record Dates: First submitted 2019-05-19; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Delirium
Keywords: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Patients with postoperative delirium.
  Interventions: Other: plasma oxidized low-density lipoprotein levels
- Control group: Patients who have not had postoperative delirium.
  Interventions: Other: plasma oxidized low-density lipoprotein levels

INTERVENTIONS:
Other: plasma oxidized low-density lipoprotein levels — Detection of plasma oxidized low-density lipoprotein levels

SUMMARY:
Postoperative delirium (POD) refers to an acute neurocognitive disorder that occurs within 1 week after surgery or before discharge. Old age is one of the important risk factors for postoperative delirium. The incidence rate of the elderly is high, and the life span of human beings is increasing. Postoperative delirium has adverse effects on both short-term and long-term outcomes, including mortality, ability to work, and dependence on society.

Low-density lipoprotein (LDL) is a key molecule in the cholesterol transport mechanism and is easily oxidized to oxidized low-density lipoprotein (OxLDL). Oxidized low density lipoproteins are immunogenic and are also cytotoxic to endothelial cells. Some studies have shown that increased oxidative stress is one of the earliest changes in disease, and similar signs can be detected in patients with Alzheimer's disease (AD) and mild cognitive impairment (MCI), such as protein oxidation and lipids. An increase in the quality of the peroxidation index. For the study of anesthesiology, oxidative stress theory has long been recognized as one of the mechanisms of postoperative delirium. We have a hypothesis that plasma oxidized low-density lipoprotein levels are associated with postoperative delirium and can be used as an early warning marker for disease occurrence.

Based on clinical research data, we conducted a prospective cohort study to explore the correlation between plasma oxidized low-density lipoprotein levels and postoperative sputum, providing clinical prediction and diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

* Surgical treatment was performed in our hospital under standard anesthesia.
* Patients in orthopedics, urology and general surgery.

Exclusion Criteria:

* Patients with mental illness or taking psychotropic substances before surgery.
* Preoperative dementia or cognitive dysfunction.
* Unable to communicate and cooperate with patients due to coma, language barrier or end-stage disease before surgery.
* ASA greater or equal to 4.
* Patients who have undergone neurosurgery and cardiac vascular surgery.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients in orthopedics, urology and general surgery .
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-20 (Estimated); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-09-20 (Estimated)

PRIMARY OUTCOMES:
plasma oxidized low-density lipoprotein levels | through study completion, an average of 4 months
  Preoperative plasma oxidized low-density lipoprotein levels
plasma oxidized low-density lipoprotein levels | through study completion, an average of 4 months
  Postoperative plasma oxidized low-density lipoprotein levels

IPD SHARING:
Plan to Share IPD: No